CLINICAL TRIAL: NCT06931405
Title: A Phase 2 Study to Evaluate the Safety, Tolerability, and Clinical Activity of BLU-808, a Wild Type KIT Inhibitor, in Chronic Inducible Urticaria and Chronic Spontaneous Urticaria
Brief Title: Study of BLU-808 in Chronic Inducible Urticaria (CIndU) and Chronic Spontaneous Urticaria (CSU)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Blueprint Medicines Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BLU-808-1201; 2024-520031-33-00 (Other: Clinical Trials Information System (CTIS))
Record Dates: First submitted 2025-04-09; First posted 2025-04-17 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Chronic Inducible Urticaria; Chronic Spontaneous Urticaria
Keywords: Chronic Inducible Urticaria; Chronic Spontaneous Urticaria; BLU-808; CIndU; CSU; Chronic Urticaria; CU; Cold Urticaria; ColdU; Symptomatic Dermographism; SD
MeSH Terms: conditions — Chronic Inducible Urticaria; Chronic Urticaria; Cold Urticaria; Familial dermographism

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Arms A1 and A3 are non-randomized and open label. Arm B is randomized and double blind.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm A1 (Part A): BLU-808 (Experimental): BLU-808 will be administered orally.
  Interventions: Drug: BLU-808
- Arm A3 (Part A): BLU-808 (Experimental): BLU-808 will be administered orally.
  Interventions: Drug: BLU-808
- Arm B (Part B): BLU-808/Placebo (Experimental): BLU-808 or matching placebo will be administered orally.
  Interventions: Drug: BLU-808; Drug: Placebo

INTERVENTIONS:
Drug: BLU-808 — Oral administration
Drug: Placebo — Oral administration
  Arms: Arm B (Part B): BLU-808/Placebo

SUMMARY:
This is a 2-part, proof-of-concept study to be conducted globally, designed to evaluate the safety, tolerability, clinical activity, pharmacokinetics, and pharmacodynamics of BLU-808, a wild type KIT inhibitor, in participants with CIndU (Part A) or CSU (Part B).

ELIGIBILITY:
Key Inclusion Criteria:

* Part A: Confirmed diagnosis of CIndU for ≥3 months prior to Day 1 that is inadequately controlled with second generation H1-antihistamines.
* Part B: Confirmed diagnosis of CSU for ≥3 months prior to Day 1 that is inadequately controlled with second generation H1-antihistamines.

Key Exclusion Criteria:

* Part A: Any active urticaria that may interfere with study assessments.
* Part B: Participant has a clearly defined predominant cause of chronic urticaria or sole trigger such as symptomatic dermographism and cold-induced urticaria.
* Part A and Part B: Any other skin disease associated with chronic itching or angioedema that might influence the study evaluations and results, skin diseases associated with only wheals and no itch, or autoinflammatory diseases with urticarial lesions.
* Part A and Part B: Significant medical, psychiatric, or surgical conditions, or physical findings that may affect participant safety, study drug metabolism, study participation, or assessment of study results.
* Part A and Part B: Abnormal laboratory values that may pose risks or interfere with study participation.
* Part A and Part B: Pregnancy or plans for pregnancy; breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2025-05-28 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Part A and Part B: Number of Participants with Treatment-emergent Adverse Events (TEAEs) | Day 1 through Week 16

SECONDARY OUTCOMES:
Part A: Mean Change From Baseline in Critical Temperature Threshold (CTT) at Week 12 | Baseline, Week 12
  CTT is the temperature at which CIndU symptoms appear.
Part A: Mean Change From Baseline in Total Fric Score (TFS) at Week 12 | Baseline, Week 12
  TFS is a measure of CIndU trigger thresholds and disease activity.
Part A and Part B: Complete Response Rate | Week 12
Part A and Part B: Absolute Change From Baseline in Serum Tryptase Concentration at Week 12 | Baseline, Week 12
Part A and Part B: Percent Change From Baseline in Serum Tryptase Concentration at Week 12 | Baseline, Week 12
Part A and Part B: Area Under the Curve (AUC) of BLU-808 | Day 1 to Day 57
Part A and Part B: Maximum Plasma Concentration (Cmax) of BLU-808 | Day 1 to Day 57
Part A and Part B: Minimum Plasma Concentration (Cmin) of BLU-808 | Day 1 to Day 57
Part A and Part B: Apparent Clearance (CL/F) of BLU-808 | Day 1 to Day 57
Part A and Part B: Apparent Volume of Distribution for the Central Compartment (Vc/F) of BLU-808 | Day 1 to Day 57
Part A and Part B: Terminal Half-life (t½) of BLU-808 | Day 1 to Day 57
Part B: Mean Change From Baseline in Urticaria Activity Score Over 7 Days (UAS7) at Week 12 | Baseline, Week 12
  UAS7 is a patient-reported outcome used to assess symptoms in participants with CSU.

CONTACTS AND LOCATIONS:
Locations (46):
- United States (26):
  - Allervie Clinical Research, Birmingham, Alabama
  - Acuro Research, Inc., Little Rock, Arkansas
  - Modena Allergy & Asthma Clinical Research - La Jolla, La Jolla, California
  - Allergy & Asthma Associates of Southern California, Laguna Niguel, California
  - Allergy & Asthma Medical Group and Research Center, San Diego, California
  - Allergy Affiliates Inc., Bradenton, Florida
  - University of South Florida, Tampa, Florida
  - Treasure Valley Medical Research, Boise, Idaho
  - Endeavor Health, Northbrook, Illinois
  - Dawes Fretzin Clinical Research Group, LLC, Indianapolis, Indiana
  - Southern Indiana Clinical Trials, New Albany, Indiana
  - The Indiana Clinical Trials Center, Plainfield, Indiana
  - Equity Medical - Bowling Green, Bowling Green, Kentucky
  - Johns Hopkins University, Baltimore, Maryland
  - Institute For Asthma & Allergy, Wheaton, Maryland
  - Chesapeake Clinical Research, White Marsh, Maryland
  - Henry Ford Health, Detroit, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - The Clinical Research Center LLC., St Louis, Missouri
  - Montana Medical Research, Inc., Missoula, Montana
  - Equity Medical (at Cameron Dermatology) - New York, New York, New York
  - Bernstein Clinical Research Center, Cincinnati, Ohio
  - Allergy & Clinical Immunology Associates, Pittsburgh, Pennsylvania
  - National Allergy, Asthma & Urticaria Centers of Charleston, Charleston, South Carolina
  - Medical University of South Carolina (MUSC), Charleston, South Carolina
  - Reveal Research Institute, Dallas, Texas
- Odense University Hospital - Odense, Odense, Denmark
- Germany (6):
  - Fraunhofer-Institut fuer Translationale Medizin und Pharmakologie ITMP - Standort Berlin, Berlin
  - Universitaetsklinikum Carl Gustav Carus Dresden, Dresden
  - Universitaetsklinikum Frankfurt - Klinikum der Johann Wolfgang Goethe Universitaet, Frankfurt am Main
  - Medizinische Hochschule Hannover (MHH), Hanover
  - Universitaetsmedizin der Johannes Gutenberg - Universitaet Mainz, Mainz
  - Universitaetsklinikum Tuebingen, Tübingen
- Italy (3):
  - Azienda Ospedale - Università Padova, Padua
  - Azienda Ospedaliero Universitaria Policlinico Umberto, Rome
  - Centro Ricerche Cliniche di Verona s.r.l., Verona
- Spain (4):
  - Hospital del Mar, Barcelona
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Universitari de Bellvitge, Barcelona
  - Hospital Regional Universitario de Malaga, Málaga
- Taiwan (6):
  - National Taiwan University Hospital Hsin-Chu Branch, Hsinchu
  - Kaohsiung Veterans General Hospital (KSVGH), Kaohsiung City
  - Taipei Medical University - Shuang Ho Hospital, New Taipei City
  - China Medical University Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Linkou Chang Gung Memorial Hospital (CGMHLK), Taoyuan